CLINICAL TRIAL: NCT02063997
Title: A Randomized, Double-Blind, Active and Placebo-Controlled Study to Evaluate the Efficacy and Safety of Arhalofenate for Preventing Flares and Reducing Serum Uric Acid in Gout Patients
Brief Title: Evaluate the Efficacy and Safety of Arhalofenate for Preventing Flares and Reducing Serum Uric Acid in Gout Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB102-21425
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — arhalofenate; Allopurinol; Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arhalofenate 600 mg (Experimental)
  Interventions: Drug: Arhalofenate 600 mg
- Arhalofenate 800 mg (Experimental)
  Interventions: Drug: Arhalofenate 800 mg
- Allopurinol 300 mg; colchicine 0.6 mg (Active Comparator)
  Interventions: Drug: Allopurinol 300 mg; Drug: Colchicine 0.6 mg
- Allopurinol 300 mg (Active Comparator)
  Interventions: Drug: Allopurinol 300 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arhalofenate 600 mg — Arhalofenate 600 mg tablets once daily for 12 weeks
  Arms: Arhalofenate 600 mg
Drug: Allopurinol 300 mg — Allopurinol 300 mg tablets once daily for 12 weeks
  Arms: Allopurinol 300 mg; Allopurinol 300 mg; colchicine 0.6 mg
Drug: Colchicine 0.6 mg — Colchicine 0.6 mg over-encapsulated tablets once daily for 12 weeks
  Arms: Allopurinol 300 mg; colchicine 0.6 mg
Drug: Placebo — Placebo tablets once daily for 12 weeks
  Arms: Placebo
Drug: Arhalofenate 800 mg — Arhalofenate 800 mg tablets once daily for 12 weeks
  Arms: Arhalofenate 800 mg

SUMMARY:
The purpose of this study is to determine whether arhalofenate is effective in preventing flares and reducing serum uric acid in gout patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 75 years of age, inclusive
* Known gout diagnosis (per criteria of the American Rheumatism Association for the classification of the acute arthritis of primary gout, see Appendix 3)
* At least three patient-reported and documented flares during the 12 months prior to screening (the first of these flares may have resulted in the gout diagnosis; any recent flare must have resolved, with the patient back to usual comfort level at least seven days prior to screening)
* Have not used any ULT since at least two weeks prior to screening
* Have not used colchicine since at least two weeks prior to screening
* Usual level of resting pain when NOT experiencing flare is three or less on an 11-point numerical rating scale (NRS)
* Have a sUA ≥ 7.5 mg/dL and ≤ 12 mg/dL at screening
* All female patients must be surgically sterile or post-menopausal (at least 45 years of age with no history of menses for at least two years); or have a partner who has undergone vasectomy or must agree to use two medically accepted methods of contraception including a barrier method (see Appendix 4) for the entire duration of study participation unless she reports complete sexual abstinence. Female patients must not be pregnant or lactating
* Estimated creatinine clearance (eCrCl) ≥ 60 ml/min/1.73m2 calculated by Cockcroft-Gault method at screening
* Liver function tests ≤ 3X ULN for AST, ALT and total bilirubin; ≤ 3X ULN for ALP and GGT; and ≤ 3X ULN for CK at screening
* All other clinical laboratory parameters must be within normal limits or considered not clinically significant
* Electrocardiogram (ECG) must be normal, or if abnormal, considered not clinically significant at screening
* Systolic blood pressure ≤ 160 mm Hg and diastolic blood pressure ≤ 90 mm Hg at screening; known hypertensive patients stable (blood pressure [BP] reading as above) with medication may be included
* Patients using agents known to influence sUA levels (see Appendix 7) must be on a stable dose and regimen for at least two weeks prior to screening and must be willing to continue the same doses and regimens during study participation
* Expected to be able to tolerate a short course of either oral NSAIDs and/or oral steroids as may be needed to treat a flare
* Must be able to swallow tablets/capsules
* Following training, must be willing and able to understand and complete an electronic diary

Exclusion Criteria:

* Receiving treatment with allopurinol, colchicine, probenecid, benzbromarone, or febuxostat within two weeks or pegloticase within six months prior to screening
* Known or suspected secondary hyperuricemia (e.g. due to myeloproliferative disorder or organ transplant)
* Diagnosis of xanthinuria
* Fractional excretion of urate > 10% at screening
* History of documented or suspected kidney stones
* Known infection with the human immunodeficiency virus (HIV) or history of viral hepatitis type B or C
* A diagnosis of illicit drug or alcohol dependence or abuse within one year of screening
* History of upper gastrointestinal (GI) bleeding, documented peptic ulcer disease (unless known H. pylori infection treated successfully without recurrence), within three years of screening
* History of stroke, transient ischemic attack (TIA), acute myocardial infarction (MI), congestive heart failure (NYHA Class II-IV), angina pectoris, coronary intervention procedure (including but not limited to angioplasty, stent placement, coronary revascularization), lower extremity bypass procedure, systemic or intracoronary fibrinolytic therapy within five years of screening
* History of cancer within five years of screening, with the following exceptions: adequately treated non-melanomatous skin cancers, non-metastatic prostate cancer or in situ cervical cancer
* Patients with a history of bladder cancer, active bladder cancer or hematuria
* Body mass index (BMI) > 42 kg/m2 at screening
* Current or expected requirement for anticoagulant therapy (except for aspirin ≤ 325 mg/day, clopidogrel [Plavix] ≤ 75 mg/day, or prasugrel [Effient] ≤ 10 mg/day)
* Use of any of the following within eight weeks prior to screening: potent CYP3A4 inhibitors, cytotoxic agents (including azathioprine, mercaptopurine, cyclosporine, cyclophosphamide, etc.), ranolazine, digoxin, theophylline, sulphonylureas, thiazolidinediones (e.g., rosiglitazone or pioglitazone), atypical antipsychotic agents, ampicillin, amoxicillin, loop diuretics or phenytoin
* Chronic treatment with NSAIDs (except for as needed [prn] use to treat acute events); per protocol a short course of oral NSAIDs may be used to treat flares during the study
* Current or expected chronic treatment with systemic corticosteroids (topical, ophthalmic, intra-articular or inhaled corticosteroid at a dose < 1600 μg/day is permitted); per protocol a short course of oral corticosteroid may be used to treat flares occurring during the study
* History of intra-articular steroid injection to treat flare within four weeks of screening
* Known hypersensitivity or intolerance to allopurinol or colchicine
* Treatment with any other investigational therapy within 30 days or within five half lives, whichever is longer, prior to screening
* Patients who received arhalofenate in a previous trial
* Any other condition(s) that would compromise the safety of the patient, prevent compliance with the study protocol including ability to use an electronic diary, or compromise the quality of the clinical study, as judged by the Investigator and/or Medical Monitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The incidence of flares (mean number of flares per patient) from baseline through Week 12 in the arhalofenate 800 mg group compared to the allopurinol 300 mg group. | 12 weeks

SECONDARY OUTCOMES:
Percent sUA reduction from baseline to Week 12 in the arhalofenate 800 mg group compared to the placebo group | 12 weeks
Percent sUA reduction from baseline to Week 12 in the arhalofenate 600 mg group compared to the placebo group | 12 weeks
Proportion of patients with sUA < 6 mg/dL at Week 12 in the arhalofenate 800 mg group compared to the placebo group | 12 weeks
The incidence of flares from baseline through Week 12 in the arhalofenate 600 mg group compared to the allopurinol 300 mg group | 12 weeks
Proportion of patients with sUA < 6 mg/dL at Week 12 in the arhalofenate 600 mg group compared to placebo group | 12 weeks
Time from baseline to onset of first flare for the arhalofenate 800 mg group compared to the allopurinol 300 mg group | 12 weeks
Time from baseline to onset of first flare for the arhalofenate 600 mg group compared to the allopurinol 300 mg group | 12 weeks

OTHER OUTCOMES:
Proportion of patients experiencing at least one flare from baseline through Week 12 | 12 weeks
Proportion of patients experiencing two or more flares from baseline through Week 12 | 12 weeks
The incidence of flares from baseline through Week 4, from Week 5 through Week 8, and from Week 9 through Week 12 | 12 weeks
Duration of flares | 12 weeks
Duration of flare treatment | 12 weeks
Flare composite score (summation of the daily maximum pain score on NRS during the duration of the flare) | 12 weeks
Proportion of patients experiencing flares who reached a sUA target < 6 mg/dL during treatment | 12 weeks
Evaluation of activity limitation associated with flare via HAQ-II | 12 weeks
Changes from baseline in fractional excretion of urate | 12 weeks
Changes from baseline in HbA1c and fasting TG in patients with HbA1c > 7.0% and TG > 150 mg/dL at baseline, respectively | 12 weeks
Adverse events (AE), and changes in vital signs and safety laboratory tests | 12 weeks
Safety-related study drug discontinuations | 12 weeks
Flare-related study drug discontinuations | 12 weeks
Steady-state arhalofenate acid serum and urine concentrations | 12 weeks

CONTACTS AND LOCATIONS:
Locations (56):
- United States (52):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - El Cajon, California
  - Long Beach, California
  - Los Angeles, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - DeLand, Florida
  - Jupiter, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Honolulu, Hawaii
  - Boise, Idaho
  - Brownsburg, Indiana
  - Bowling Green, Kentucky
  - Elizabethtown, Kentucky
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Hagerstown, Maryland
  - Olive Branch, Mississippi
  - St Louis, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Brooklyn, New York
  - New York, New York
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Johnstown, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Greer, South Carolina
  - Summerville, South Carolina
  - Bristol, Tennessee
  - Jackson, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Spokane, Washington
  - Clarksburg, West Virginia
- Canada (3):
  - Newmarket, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
- Tbilisi, Georgia

REFERENCES:
- [Derived] Poiley J, Steinberg AS, Choi YJ, Davis CS, Martin RL, McWherter CA, Boudes PF; Arhalofenate Flare Study Investigators. A Randomized, Double-Blind, Active- and Placebo-Controlled Efficacy and Safety Study of Arhalofenate for Reducing Flare in Patients With Gout. Arthritis Rheumatol. 2016 Aug;68(8):2027-34. doi: 10.1002/art.39684. PMID 26989892